CLINICAL TRIAL: NCT02479997
Title: Clinical Application of Dual Sentinel Lymph Node Staining Method in Breast Cancer Patients Who Receive Neoadjuvant Therapy(Chemotherapy, Hormonal Therapy, Targeted Therapy); Clinical Study for 130 Patients
Brief Title: Clinical Application of Dual Sentinel Lymph Node Staining Method in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Seeyoun Lee, Medical Doctor, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NCC-1410201-2
Record Dates: First submitted 2015-05-08; First posted 2015-06-24 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant chemotherapy; Indocyanine green (ICG); Radioisotope (RI); Near infrared fluorescence camera
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green; Radioisotopes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radioisotope (RI) (Active Comparator): Using RI only as SLNB mapping in breast cancer patients who receive neoadjuvant chemotherapy.
  Interventions - patient assigend RI groups are injected only RI
  * fill the Primay Case Report Form during surgery
    * PCRF including SLN detection time, duration of SLN approch time to 1st sentinel node dection time, incision length , depth, RI +/- .
  Interventions: Drug: Indocyanine green; Drug: Radioisotope
- Indocyanine green (ICG) +RI (Active Comparator): Dual sentinel node staining method using mixture of indocyanine green (ICG) and radioisotope (RI) in breast cancer patients who receive neoadjuvant chemotherapy.
  Interventions - patient assigend RI groups are injected RI +ICG
  * prepare fluorescence camera when the surgery begin
  * surgeon uses the camera to decect fluorescence flow on SLN
  * fill the Primay Case Report Form during surgery
    * PCRF including SLN detection time, duration of SLN approch time to 1st sentinel node dection time, incision length , depth, RI +/- , ICG+/-
  Interventions: Drug: Indocyanine green; Drug: Radioisotope

INTERVENTIONS:
Drug: Indocyanine green — ICG is cyanine dye used in medical diagnostics. It is used for determining cardiac output, hepatic function, and liver blood flow, and for ophthalmic angiography.
  In this study, Investigator uses ICG as a fluorescent dye which is used in medicine as an indicator substance . And it will allow detection of SLN more convenientlty.
  Other Names: ICG
Drug: Radioisotope — Nuclear medicine uses radiation to provide diagnostic information about the functioning of a person's specific organs, or to treat them. Diagnostic procedures using radioisotopes are now routine.
  Other Names: RI

SUMMARY:
This study aimed to compare detection rate between dual sentinel node staining method using mixture of indocyanine green (ICG) with radioisotope(RI), and RI only.

To identify the first lymph node(s) along the lymphatic drainage pathway from the primary tumor in the breast cancer using RI only has several disadvantages such as invisibility, interference. As ICG can be visualized with a fluorescence imaging system, we expects dual sentinel lymph node staining method had better outcomes.

DETAILED DESCRIPTION:
Using mixture of indocyanine green (ICG) with radioisotope (RI) can guide surgeons to identify the first lymph node(s) along the lymphatic drainage pathway from the primary tumor in the breast to the axillary lymph node basin.

Last pilot study, sentinel lymph node was successfully identified by using dual method of ICG and RI in 5 patients. In this study, when radiolabeled colloid is used, a gamma probe identifies radioactivity in the lymph nodes in the axilla. If ICG, RI both used, Near infrared fluorescence camera visualized during surgery.

As investigators measure node detection time from axillary approach moment, investigators are going to compare detection rate. (ICG+RI or RI only). And determine the accuracy.

Sentinel lymph node mapping with both ICG and radiolabeled colloid mapping agents was recommended to maximize the likelihood of SLN identification and to minimize the possibility of missing SLNs, which could result in a false-negative event.The protocol required that 130 patients who receive neoadjuvant chemotherapy.

In this study investigators expects using mixture of indocyanine green (ICG) with radioisotope (RI) has potential to improve sentinel lymph node (SLN) mapping in breast cancer patients who receive neoadjuvant chemotherapy.

Sentinel lymph node mapping with both ICG and radiolabeled colloid mapping agents was recommended to maximize the likelihood of SLN identification and to minimize the possibility of missing SLNs, which could result in a false-negative event.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients who receive neoadjuvant therapy (chemotherapy,hormonal therapy, targeted therapy)
* cN1-cN2 or cN3( but must be complete response status)on tumor lymphnode metastasis classification( TNM) after neoadjuvant therapy.
* ECOG Performance status 0 or 1
* consented patients with more than 20 years, less than 70 years

Exclusion Criteria:

* history of breast cancer
* early stage breast cancer
* history of excisional or incisional biopsy or axillary dissection
* inflammatory breast carcinoma
* cN3 on tumor lymphnode metastasis classification(TNM)
* stage 4 breast cancer
* pregnancy

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Identification rate of sentinel lymphnode biopsy | Participants will be followed for 2 weeks from operation

SECONDARY OUTCOMES:
Duration of sentinel lymphnode biopsy | 3months follow up from the day of operation

CONTACTS AND LOCATIONS:
Overall Officials: Seeyoun Lee, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea